CLINICAL TRIAL: NCT01249950
Title: Study on the Appropriateness of Bariatric Surgery in Adolescents
Status: Terminated | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 08 157 02; 2008-A01320-55 (Other: AFSSAPS)
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2013-11-11 (Estimated); Status verified 2013-11

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; teenagers; co-morbidities; bariatric surgery; epidemiology
MeSH Terms: conditions — Obesity, Morbid | interventions — Feasibility Studies

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adolescents: adolescents with morbid obesity
  Interventions: Other: feasibility

INTERVENTIONS:
Other: feasibility — feasibility

SUMMARY:
single-center study carried out in order to evaluate in prospective among patients seen or treated in the pediatric endocrinology unit and multidisciplinary management of obesity, the potential number of patients eligible for surgery.

DETAILED DESCRIPTION:
This is a feasibility study in order to file a subsequent national project as part of a PHRC on bariatric surgery in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* failure of weight loss in an organized care> 6 months
* BMI > à 35 kg/m2 with presence of severe co-morbidities (diabetes, moderate or severe OSAS, intracranial hypertension, severe hepatic steatosis), which can be improved by a significant weight loss and sustainable OR BMI > or = 40 kg/m2 with less severe co-morbidities (hypertension, GERD) and may worsen the health status including reduced quality of life.
* Patients must have completed their growth (bone age > 13 for girls and >15 for boys).
* The teenager and his legal representative must have given their informed consent.
* The subject must be affiliated to a social security scheme

Exclusion Criteria:

* syndromic obesities
* tumor-induced obesity
* Patient with severe psychiatric disorders
* Patient with eating disorders
* Patients under judicial protection
* Patient under guardianship or curatorship
* Patient participating in another study

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: adolescents
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-10; Primary Completion 2011-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
potential number of patients eligible for surgery | 24 months
  evaluate prospectively the potential number of patients eligible for surgery, among patients seen or treated in the pediatric endocrinology unit and multidisciplinary management of obesity.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice JOURET, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse, France